CLINICAL TRIAL: NCT06679218
Title: Improving Health Status in COVID-19 Long-Hauler Through an Activity Coaching Programme: a Randomized Control Trial
Brief Title: Improving Health Status in COVID-19 Long-Hauler
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, Principal Investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DF0102UG
Record Dates: First submitted 2024-11-06; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Post COVID-19 Condition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Activity Coaching Programme (Experimental)
  Interventions: Other: Activity Coaching Programme
- Standard medical care and leaflet education (Active Comparator)
  Interventions: Other: Standard medical care and leaflet education

INTERVENTIONS:
Other: Activity Coaching Programme — The intervention will consist of individualized physical activity coaching sessions, which will take place twice a week for 8 weeks. These sessions will focus on encouraging progressive and personalized physical activity according to each participant's ability. The sessions will also include relaxation techniques, targeted ventilation and strategies to improve activity management.
  Arms: Activity Coaching Programme
Other: Standard medical care and leaflet education — In addition to standard medical care, patients assigned to this group received a leaflet with information about the main post COVID-19 condition symptoms. This is a control group that was not controlled or monitored by a therapist.
  Arms: Standard medical care and leaflet education

SUMMARY:
This randomized clinical trial investigates the effects of a distance physical activity coaching program on the health of COVID-19 long-hauler. The study evaluates the impact of individualized coaching interventions to improve participants' physical activity and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes.
* Agreed to participate.
* Post COVID-19 condition patients meeting the WHO definition for this disease.
* Sedentary patients according to the cut-off point of the International Physical Activity Questionnaire (IPAQ).

Exclusion Criteria:

* Pulmonary, cardiac, neurological, vascular, or orthopaedic pathologies that could limit the execution of the evaluation and intervention.
* Cognitive impairment that prevented them from understanding and answering the questionnaires.
* Patients suffering from a reinfection with SARS-CoV-2.
* Patients with a history of severe or critical COVID-19 disease severity.
* Patients participating in other studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-11 (Estimated); Primary Completion 2025-01-11 (Estimated); Study Completion 2025-01-20 (Estimated)

PRIMARY OUTCOMES:
IPAQ (International Physical Activity Questionnaire) | Baseline and at 8 weeks at the end of the intervention
EQ-5D (EuroQol-5 Dimensions) | Baseline and at 8 weeks at the end of the intervention
PROMIS (Patient-Reported Outcomes Measurement Information System) | Baseline and at 8 weeks at the end of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Marie Carmen Valenza, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- Faculty of Health Sciences. University of Granada, Granada, Granada, Spain